CLINICAL TRIAL: NCT06816680
Title: Comparison of Keratinized Mucosa Width Increase Around Implants Between Palatal Pedicle Flap and Free Gingival Graft: a Clinical Controlled Trial
Brief Title: Comparison Between Free Gingival Graft and Palatal Pedicle Flap
Acronym: Pedicle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202100738A3D001
Record Dates: First submitted 2025-01-19; First posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-01

CONDITIONS: Peri-Implant Health; Peri-Implant Tissues; Peri-implant Bone Level
Keywords: Mucogingival Surgery; Dental Implants; Keratinized Tissue; Soft Tissue Augmentation; Free Gingival Graft; Pedicle Graft
MeSH Terms: interventions — fibrinopeptides gamma

STUDY DESIGN:
Intervention Model Description: Patients requiring KMW gain during uncovering surgery were included. Two surgical methods were compared: apically position flap with free gingival graft (FGG group) and the palatal pedicle flap with collagen matrix (PPF group). The primary outcomes were KMW amount and shrinkage rate at 2 weeks (2W) and 2 months (2M), 3 months (3ML), and 6 months after loading (6ML). Secondary outcomes included the intra- and inter- group comparison in mucosal recession (REC), probing pocket depth (PPD), marginal bone level (MBL) and restoration designs.
Who Masked: Participant, Outcomes Assessor
Masking Description: Patient did not know which intervention was performed, and the independent assessor of radiographic films was blinded to which intervention was done either.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- FGG group (Active Comparator): In APF + FGG technique, a split- thickness flap was prepared and apically positioned using 5-0 (PDS*II, Polydioxanone, ETHICON) or 6-0 (PROLENE, ETHICON) sutures for flap stabilization.
  Interventions: Procedure: APF + FGG
- Palatal pedicle flap with collagen matrix (Active Comparator): For thepalatal pedicle flap with collagen matrix (PPF) group, the palatal sliding flap was a modified version of modified roll technique, the crestal incision was placed 5 mm palatally from the border of keratinized tissue to allow for KMW redistribution, and a partially split-thickness flap was harvested from palatal connective tissue graft (CTG).
  Interventions: Procedure: PPF group

INTERVENTIONS:
Procedure: APF + FGG — In APF + FGG technique, a split- thickness flap was prepared and apically positioned using 5-0 (PDS*II, Polydioxanone, ETHICON) or 6-0 (PROLENE, ETHICON) sutures for flap stabilization. To eliminate muscle and frenum attachment at recipient site, vestibuloplasty and a periosteal incision were performed. A 4 mm or 6 mm healing abutment was then screwed onto the implants. FGG was harvested from palate in a 7-8 mm width and trimmed to an even thickness of 1 to 1.5 mm. A resorbable hemostatic sponge (Spongostan, Ethicon, Johnson & Johnson) was placed at donor site for wound coverage. For graft fixation, a loop suture with 6-0 (PROLENE, ETHICON) was first placed at the center of recipient site, additional sutures were added to enhance stabilization.
  Other Names: free gingival graft
  Arms: FGG group
Procedure: PPF group — For the PPF group, the palatal sliding flap was a modified version of modified roll technique, as described in previous cohort study. Unlike the original technique, the crestal incision was placed 5 mm palatally from the border of keratinized tissue to allow for KMW redistribution, and a partially split-thickness flap was harvested from palatal connective tissue graft (CTG). Following buccal pouch flap preparation, a slight APF was required in cases with limited vestibular depth. When the palatal pedicle CTG was rolled in buccal pouch flap, a loop suture with 6-0 (PROLENE, ETHICON) was used for flap stabilization.
  Other Names: palatal pedical flap
  Arms: Palatal pedicle flap with collagen matrix

SUMMARY:
Patients requiring KMW gain(mm) during uncovering surgery were included. Two surgical methods were compared: apically position flap with free gingival graft (FGG group) and the palatal pedicle flap with collagen matrix (PPF group). The primary outcomes were KMW amount(mm) and shrinkage rate(%) at 2 weeks (2W) and 2 months (2M), 3 months (3ML), and 6 months after loading (6ML). Secondary outcomes included the intra- and inter- group comparison in mucosal recession (REC, mm), probing pocket depth (PPD, mm), marginal bone level (MBL, mm) and restoration designs.

DETAILED DESCRIPTION:
The present prospective clinical controlled trial included patients with at least one implant requiring stage 2 surgery. All implant surgeries were performed by the same surgeon (CYL) from 2021 July to 2023 January. All included patients had to meet the following inclusion criteria:

1. Patient had at least one bone-level 3i implant*: 3.25, 4, and 5 mm in diameter, 8.5, 10, and 11.5 mm in length, and primary stability with an insertion torque ≥ 20Ncm. All implants needed to be free of peri-implant disease.
2. Informed consent had been obtained prior to implant uncovering.
3. Insufficient keratinized mucosal width (KMW< 2mm) was observed
4. Complete data, including both clinical and radiographic outcomes, was available
5. The patient followed the supportive postimplant regimen for a 12-month loading period, indicating good compliance.

Patients were excluded from this project if they have one of the following conditions:

1. Untreated periodontitis.
2. Uncontrolled systemic disease, such as hypertension, diabetes, and heavy smokers (more than 10 pieces per day).
3. History of radiation therapy on head and neck regions.
4. Patient with pregnancy
5. Patient had pathologic lesions around peri-implant mucosa
6. Guided bone regeneration was needed concomitantly with soft tissue phenotype modification during uncovering surgery.

Following the revised version of Helsinki Declaration in 2013, the protocol of current trial was conducted and approved by institutional review board of Chang Gung memorial hospital (IRB: 202100738A3). The cohort study was performed in accordance with STROBE statement.

2.2 Clinical Procedures Under local anesthesia, either APF combined with FGG or PPF with xenogenic matrix was performed around implants for KMW enhancement, which was concomitant with uncovering surgery.

In APF + FGG technique, a split- thickness flap was prepared and apically positioned using 5-0 (PDS*II, Polydioxanone, ETHICON) or 6-0 (PROLENE, ETHICON) sutures for flap stabilization. To eliminate muscle and frenum attachment at recipient site, vestibuloplasty and a periosteal incision were performed. A 4 mm or 6 mm healing abutment was then screwed onto the implants. FGG was harvested from palate in a 7-8 mm width and trimmed to an even thickness of 1 to 1.5 mm. A resorbable hemostatic sponge (Spongostan, Ethicon, Johnson & Johnson) was placed at donor site for wound coverage. For graft fixation, a loop suture with 6-0 (PROLENE, ETHICON) was first placed at the center of recipient site, additional sutures were added to enhance stabilization.

For the PPF group, the palatal sliding flap was a modified version of modified roll technique, as described in previous cohort study. Unlike the original technique, the crestal incision was placed 5 mm palatally from the border of keratinized tissue to allow for KMW redistribution, and a partially split-thickness flap was harvested from palatal connective tissue graft (CTG). Following buccal pouch flap preparation, a slight APF was required in cases with limited vestibular depth. When the palatal pedicle CTG was rolled in buccal pouch flap, a loop suture with 6-0 (PROLENE, ETHICON) was used for flap stabilization. The exposed connective tissue bed or bone around the implants was covered with a dual- layered collagen matrix (Lyoplant®Onlay, Aesculap), and additional sutures were used for graft and flap fixation. The specific indications for the PPF technique were shown as below: (1) the total keratinized mucosa width should be more than 3 mm; (2) the vertical soft tissue height should be more than 2 mm at the time of the uncovering surgery.

Post-operative instructions were instructed individually, and the medications were prescribed (acetaminophen 500 mg, tid for 5 days; amoxicillin 375 mg, tid for 5 days) for pain and infection control during post-operative phase. Two weeks after surgery, sutures were removed, and surgical wounds were followed at recall visit 2 months later. The implant prosthesis was then restored by prosthodontic specialists. The clinical and radiographic data were collected at 3, 6, and 12 months after loading during a strict maintenance period, which involved a 3-month interval over the course of 12 months. According to the supportive strategy, routine coronal prophylaxis with ultrasonic device and titanium curettes was applied, and oral hygiene reinforcement with adequately interdental brush and superfloss was instructed at every visit.

ELIGIBILITY:
Inclusion Criteria:

1. Patient had at least one bone-level 3i implant*: 3.25, 4, and 5 mm in diameter, 8.5, 10, and 11.5 mm in length, and primary stability with an insertion torque ≥ 20Ncm. All implants needed to be free of peri-implant disease.
2. Informed consent had been obtained prior to implant uncovering.
3. Insufficient keratinized mucosal width (KMW< 2mm) was observed
4. Complete data, including both clinical and radiographic outcomes, was available
5. The patient followed the supportive postimplant regimen for a 12-month loading period, indicating good compliance.

Exclusion Criteria:

1. Untreated periodontitis.
2. Uncontrolled systemic disease, such as hypertension, diabetes, and heavy smokers (more than 10 pieces per day).
3. History of radiation therapy on head and neck regions.
4. Patient with pregnancy
5. Patient had pathologic lesions around peri-implant mucosa
6. Guided bone regeneration was needed concomitantly with soft tissue phenotype modification during uncovering surgery.

Ages: 47 Years to 71 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-06-27 (Actual); Primary Completion 2022-06-23 (Actual); Study Completion 2023-03-07 (Actual)

PRIMARY OUTCOMES:
Keratinized mucosal width amount(mm) | at 2 weeks (2W) and 2 months (2M), 3 months (3ML), and 6 months after loading (6ML)
  Keratinized mucosal width amount(mm) was measured with periodontal probe from mucosal margin to mucosogingival junction

SECONDARY OUTCOMES:
Mucosal recession (REC, mm) | at 2 months (2M), 3 months (3ML), and 6 months after loading (6ML)
  The distance from abutment top to mucosal margin

OTHER OUTCOMES:
Probing pocket depth (PPD, mm) | 2 months(2M), 3- and 6- month loading(3ML, 6ML)
  the pocket depth was measured with periodontal probe at 6 points around the implants
Marginal bone level (MBL, mm) | 3-month and 6 month loading(3ML, 6ML)
  The distance from bone-implant contact to platform of the implant was evaluated ion peri-apical film
Emergence profile | 3- month loading
  The 3 restoration categories with straight, concave and convex.
Emergence angle (degree) | 3- month loading
  the angle between the profile and long axis of implant

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Chang Gung Memorial hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
The data that support the findings of this study are available from the corresponding author upon request.